CLINICAL TRIAL: NCT00185835
Title: Phase I Study of Cisplatin And ZD1839 (IRESSA®) in Combination With Concomitant Re-Irradiation in Patients With Loco-Regional Recurrent Squamous Cell Cancer of the Head and Neck
Brief Title: Cisplatin and ZD1839 + Re-Irradiation in Recurrent Squamous Cell Cancer of the Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: American Society of Clinical Oncology (Other); AstraZeneca (Industry)
Responsible Party: Quynh-Thu Le, Stanford University School of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ENT0012; ENT0012; NCT00185835
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2010-03-29 (Estimated); Status verified 2010-03

CONDITIONS: Head and Neck Cancer; Carcinoma, Squamous Cell
MeSH Terms: conditions — Head and Neck Neoplasms; Carcinoma, Squamous Cell | interventions — Gefitinib; Cisplatin

INTERVENTIONS:
Drug: ZD-1839
Drug: Cisplatin

SUMMARY:
To determine safety profile of the epidermal growth factor receptor (EGFR) antagonist, ZD1839 in combination with cisplatin and radiation therapy in patients with local-regional recurrent squamous cell cancer of the head and neck.

To study the effects of ZD1839 combined with either cisplatin or radiotherapy on signal transduction pathway gene expression in tumor cells in patients with local-regional recurrent squamous cell cancer of the head and neck using micro array analysis from tumor samples taken at the time of relapse and during treatment.

ELIGIBILITY:
Inclusion Criteria:- Patients must have pathologically confirmed recurrence (reappearance of previously cleared) squamous cell cancer primary in the upper aerodigestive tract or a second squamous cell primary (excluding nasopharynx or salivary gland tumors). Patients may have experienced more than one recurrence as long as the first recurrence occurred greater than or equal to 6 months following the end of the prior RT.

* The recurrence or second primary must have defined bi- or uni-dimensional measurements.
* Recurrence or second primary must be confined to the head and neck above the clavicles (loco-regional recurrence).
* The patient must not be a candidate for complete surgical resection. The previous irradiation must not exceed a maximum of 75 Gy.
* The entire tumor volume must be included in a treatment field that limits the total spinal cord dose to 50 Gy (prior RT and anticipated RT).
* Patients must be at least 6 months from prior radiation therapy.
* Patients may have received prior chemotherapy as a component of their primary treatment, but not for recurrent disease.
* Zubrod performance status 0-1.
* Granulocytes greater than or equal to 1500/mm3, platelets greater than or equal to 100,000/mm3, serum bilirubin less than or equal to 1.5 mg/dl, creatinine less than or equal to 1.5 mg/dl within 2 weeks prior to registration.
* LFT's less than or equal to 2 x normal (SGOT/SGPT/Alkaline Phosphatase). If greater than 2 x normal, liver ultrasound or CT is required to exclude metastases. If negative for metastases, patients are eligible.
* Must be able to submit previous radiation records, including simulation and portal films, in order to assure that cord tolerance is not exceeded.
* Patients must sign a study-specific informed consent form prior to study entry. Exclusion Criteria:- Primary in the nasopharynx or the salivary gland.
* Intercurrent medical illnesses which would impair patient tolerance to therapy or limit survival.
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to ZD1839 or other agents used in study.
* Pregnant and nursing women are excluded because of the potential teratogenic effects and potential unknown effects on nursing newborns.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2002-06; Primary Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
To determine safety profile of the epidermal growth factor receptor (EGFR) antagonist, ZD 1839 in combination with cisplatin and radiation therapy in patients with local-regional recurrent squamous cell cancer of the head and neck | no known

SECONDARY OUTCOMES:
To estimate the median and one-year disease-free and overall survival rates of the treated patients. | one year
To determine the response rate, duration of response and duration of stable disease in these treated patients.
To identify and estimate the incidence rate of acute and late toxicities associated with combined ZD1839, chemotherapy and re-irradiation in patients with recurrent squamous cell cancer of the head and neck. | no known
To determine the pattern of disease progression in recurrent disease patients treated with this regimen.
To assay EGFR pathway-related proteins by IHC and cDNA microarray, and to correlate their baseline expression, as well as changes in expression after therapy, with clinical endpoints including tumor remission and one-year survival. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Quynh-Thu Le, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States